CLINICAL TRIAL: NCT04038138
Title: Clinical Trial Readiness Network FSHD France: Prospective 24 Months MRI Study
Acronym: ReSOLVE_France
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-PP-04
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Muscular Dystrophy; Facioscapulohumeral
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with facioscapulohumeral muscular dystrophy (Experimental)
  Interventions: Diagnostic Test: Validation of new COA for FSHD patients

INTERVENTIONS:
Diagnostic Test: Validation of new COA for FSHD patients — Monitoring of commonly used and news COA in patients with facioscapulohumeral muscular dystrophy

SUMMARY:
The overall aim of this study is to hasten drug development for facioscapulohumeral muscular dystrophy (FSHD). Recent breakthroughs in FSHD research have identified the primary disease mechanism as the aberrant expression of a normally silenced gene, DUX4, resulting in a toxic gain-of-function. This disease mechanism is particularly amenable to knock-down of DUX4 using epigenetic strategies or RNA therapies, as well as to other interventions targeting the downstream effects of DUX4 expression. There are many drug companies actively working towards disease-targeted therapies, and two clinical trials either under way now, or planned to start in early Fall 2016. However, meetings with industry, advocacy groups, and FSHD researchers have identified several gaps in the clinical trial arsenal, and clinical trial planning as a major goal for the community. Consequently, there is an urgent need to establish the tools necessary for the conduct of currently planned and expected therapeutic trials in FSHD.

To this end, the researchers propose to develop two novel clinical outcome assessments (COA), a composite functional outcome measure (FSH-COM) and skeletal muscle biomarker, electrical impedance myography (EIM). In addition there is broad consensus a better understanding of the relationship of genetic and demographic features to disease progression will be necessary for enumerating eligibility criteria.

The specific aims are to: 1. Determine the multi-site validity of the COAs, 2. Compare the responsiveness of new COAs to other FSHD outcomes and determine the minimal clinically meaningful changes, and 3. establish FSHD cohort characteristics useful for determining clinical trial eligibility criteria. To achieve these aims, the Nice University Hospital is conducting a monocentric, prospective, 18 month study on 30 subjects.

ELIGIBILITY:
Inclusion Criteria

* Genetically confirmed FSHD1 or clinical diagnosis of FSHD with characteristic findings on exam and an affected parent or offspring 63
* Age 18-75 years
* Symptomatic limb weakness
* Patient able to walk alone or with a walking aid.
* Manual Muscle Testing (MMT) score ≥ 4 for one of the lower limb muscles
* Patient affiliated to the social security system
* Patient giving written consent after written and oral information.
* If taking over the counter supplements willing to remain consistent with supplement regimen throughout the course of the study

Exclusion Criteria

* Cardiac or respiratory dysfunction (deemed clinically unstable, or would interfere with safe testing in the opinion of the Investigator)
* Orthopedic conditions that preclude safe testing of muscle function
* Regular use of available muscle anabolic/catabolic agents such as corticosteroids, oral testosterone or derivatives, or oral beta agonists
* Use of an experimental drug in an FSHD clinical trial within the past 30 days
* Pregnancy.
* Contraindication for muscle MRI
* Any major comorbidity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
Validate FSHD-COM in French as COA | at baseline, 12, 18 and 24 months
  The FSHD-COM is an 18-item evaluator-administered instrument comprised of individually validated functional motor tasks. The body regions represented match areas of importance identified by patients and include: leg function; shoulder and arm function; trunk function, hand function; and balance. Each item is scored on a 0-4 scale, with 0 representing unaffected/normal performance, and the divisions based on healthy population normative values, or the relative degree of ability to perform the functional task. The total scale has 72 points, with larger weight given to the two most frequently patient-cited areas of functional motor concern - leg function and shoulder and arm function.
Validate optimized Timed Up and Go Test (optimized TUG) as COA | at baseline, 12, 18 and 24 months
  Balance and mobility in patients able to walk at most 30 meters will be assessed using the optimized Timed Up and Go test (TUG). The optimized TUG test measures, in seconds, the time taken by patient to sit up from a lying down position (1st time interval); stand up from the mat (approximate height of 46 cm, walk 3 meters, turn, walk back to the mat, sit down (2nd time interval); and lie down to return to starting position (3rd time interval).

SECONDARY OUTCOMES:
Change of the Motor Function Measure-32 (MFM-32) from Baseline to 12, 18 and 24 months | at baseline, 12, 18 and 24 months
  Within MFM-32, 32 terms will be evaluated to describe patient's motor functions and grouped into 3 sub-scores at baseline, 6, 12 and 24 months:
  D1: standing position and transfer D2: axial and proximal motor function D3: distal motor function The MFM-32 ratings rely on the use of a 4-point Likert scale based on the subject's maximal abilities without assistance (0: cannot initiate the task or maintain the starting position; 1: performs the task partially; 2: performs the task incompletely or imperfectly; 3: performs the task fully and normally.)
Validate the Severity Scores (CSS) as COA | at baseline, 12, 18 and 24 months
  A limited physical exam and strength testing will be used to derive a FSHD clinical severity score. The severity score ranks weakness in the face, shoulders, arms, distal, and proximal lower extremities on a 10 point scale.
Validate the Severity Scores (FCS) as COA | at baseline, 12, 18 and 24 months
  A limited physical exam and strength testing will be used to derive a FSHD clinical severity score. The severity score ranks weakness in the face, shoulders, arms, distal, and proximal lower extremities on a 15 point scale.
Change of the Manual Muscle Testing (MMT) from Baseline to 12, 18 and 24 months | at baseline, 12, 18 and 24 months
  The Manual Muscle Testing is a modified Medical Research Council 13-point and is used with standardized positions for each grade and each muscle following the recommendations of the FSH-DY Group. Shoulder abduction and flexion, elbow flexion and extension, wrist flexion and extension, fingers flexion and extension, hip flexion and abd/adduction, knee flexion and extension, ankle plantarflexion and dorsiflexion strength will be measured bilaterally
Validate the Quantitative Muscle Testing (QMT) as COA | at baseline, 12, 18 and 24 months
  Quantitative Muscle Assessment is performed using a fixed myometry testing system, with a force transducer attached by an inelastic strap to a metal frame.
Validate the fall and exercice questionnaire as COA | at baseline, 12, 18 and 24 months
  A fall and exercise questionnaire will assess average monthly falls and near falls, and average weekly amount of exercise. A fall assessment will be completed weekly for 3 months after the first visit. Subjects will be asked to respond to a call every week, for 12 consecutive weeks, that asks about any falls they have had over the past week.
Validate the work questionnaire as COA | at baseline, 12, 18 and 24 months
  The work questionnaire is a standard questionnaire asking about the effect of FSHD on work/occupation.
Validate the Patient-Reported Outcomes Measurement Information System-57 (PROMIS57) as COA | at baseline, 18 and 24 months
  The PROMIS57 is an instrument developed by the NIH PROMIS initiative. It generates scores for physical function, and the impact of physical limitations on daily life.
Validate the Upper Extremity Functional Index 15 (UEFI15) as COA | at baseline, 18 and 24 months
  The Upper Extremity Functional Index 15 (UEFI15) is a validated patient reported measure for adults with upper extremity dysfunction. This index measures upper extremity dysfunction. 20 questions are combined into a total score, the score is transformed into a normalized score with 80 representing normal, and lower scores representing increasing disability.
Validate the Facial Disability Index (FDI) as COA | at baseline, 18 and 24 months
  The Facial Disability Index (FDI) is a short 5 items questionnaire which assesses the physical impact of facial weakness. The five questions are summed into total score which transformed onto a percentage scale, with 100 representing normal, and lower scores representing increasing disability.
Validate the Iowa Oral Performance Instrument (IOPI) as COA | at baseline, 12, 18 and 24 months
  IOPI is a means to quantify lip, tongue, and buccal strength using a validated tool with published ranges for normative data for lingual measurements.
Validate Muscle Magnetic Resonance Imaging (MRI) as COA | at baseline, 12 and 24 months
  Muscle MRI studies will be performed on a 1.5 Tesla equipment at baseline,12 and 24 months
Change of the respiratory function (sitting and bedside spirometry) from Baseline to 12, 18 and months | at baseline, 12, 18 and 24 months
  Sitting and bedside spirometry allow to obtain forced vital capacity and forced respiratory volume in 1 second, two standardized outcomes commonly used to evaluate respiratory function in clinical follow up and clinical trials.
Validate the Sydney Swallow Questionnaire (SSQ) as COA | at baseline, 18 and 24 months
  The Sydney Swallow Questionnaire (SSQ) is a 17 question, self-report inventory, which was developed to measure symptomatic severity of oral-pharyngeal dysphagia as reported by the affected patient. The questionnaire uses a 100mm long visual analogue scale (VAS) for all but one question.
Validate the Multidimensional Dyspnea Profile (MDP) as COA | at baseline, 18 and 24 months
  The Multidimensional Dyspnea Profile (MDP) is a questionnaire which assesses overall breathing discomfort, sensory qualities, and emotional responses in laboratory and clinical settings. The MDP assesses dyspnea during a specific time or a particular activity (focus period) and is designed to examine individual items that are theoretically aligned with separate mechanisms.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHRU de Lille, Lille, Hauts-de-France
  - CHU de Nice, Nice, Provence-Alpes-Côte d'Azur Region
  - Myology institute Association, Paris, Île-de-France Region